CLINICAL TRIAL: NCT04281186
Title: Retinal and Cognitive Dysfunction in Type 2 Diabetes: Unraveling the Common Pathways and Identification of Patients at Risk of Dementia
Brief Title: Retinal and Cognitive Dysfunction in Type 2 Diabetes
Acronym: RECOGNISED
Status: Completed | Type: Observational
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Queen's University, Belfast (Other); Association for Innovation and Biomedical Research on Light and Image (Other); UMC Utrecht (Other); University of Medical Centre Amsterdam (Unknown); University of Rome Tor Vergata (Other); Ospedale San Raffaele (Other); University of Milan (Other); University of Southern Denmark (Other); Azienda Ospedaliero Universitaria Maggiore della Carita (Other); Hospital Mutua de Terrassa (Other); Institut Catala de Salut (Other Government); University of Montenegro (Other); Clinical Center of Montenegro (Other); University of Cadiz (Other); European Infrastructure for Translational Research (Unknown); Alzheimer Europe (Other); International Diabetes Federation Europe (Unknown); Anaxomics Biotech S.L. (Unknown); Oxurion (Industry); Genesis Biomed (Unknown)
Responsible Party: Principal Investigator, Andreea Ciudin, Prof. Dr. Rafael Simo Canonge, Hospital Universitari Vall d'Hebron Research Institute
Other Study IDs: ECR-RET-2019-14
Record Dates: First submitted 2020-02-18; First posted 2020-02-24 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Retinal Function; Cognitive Dysfunction; Microperimetry
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cross-sectional cohort: Up to 720 type 2 diabetic patients (>5 years duration), older than 65 years of age are expected to be recruited in orfer to asure the sample of 168 patients with MCI and 63 normocognitive fulfilling criteria for the prospective study.
- Prospective study-MCI: Target 168 Patients from the cross-sectional cohort diagnosed with mild cognitive impairment during the cross-sectional evaluation
- Prospective study normocognitive: 63 Patients from the cross-sectional cohort without mild cognitive impairment evaluated during the cross-sectional evaluation

SUMMARY:
The retina shares similar embryologic origin, anatomical features and physiological properties with the brain and hence offers a unique and accessible "window" to study the correlates and consequences of subclinical pathology in patients with cognitive impairment. Our hypothesis is that the neurodegeneration of the retina will run in parallel to the neurodegeneration of the brain and, therefore, the signs of neurodysfunction in the retinal assessment will be more evident in those patients with rapid cognitive decline. Microangiopathy will also participate in cognitive decline and its specific role, as well as usefulness of retinal imaging, will be also examined.

This is a multinational and multicentre cross-sectional study and prospective, longitudinal cohort observational study.

DETAILED DESCRIPTION:
The study consists of two main parts: a cross-sectional part and a longitudinal part, aimed at a) to determine whether functional and/or structural retinal biomarkers or circulating biomarkers are able to differentiate people with mild cognitive impairment (MCI) within the type 2 diabetes (T2D) population (the investigators will be able to do in the cross-sectional study, and, thus, use retina and/or blood biomarkers as a potential proxy to events taking place in the brain); b)to determine whether functional and/or structural retinal biomarkers or circulating biomarkers can be used to determine the speed of cognitive decline in people with T2D and MCI and those at higher risk of developing dementia.

The cross-sectional study will allow characterization of a large group of individuals with T2D (720 participants) and establish correlations between the various functional and structural retinal endpoints obtained and the presence/absence of mild cognitive impairment (MCI) and dementia. The cross-sectional study will allow identification of T2D patients with MCI; of these a group of 168 T2D patients with MCI and a group of T2D patients without MCI (n=63), which will act as a control group, will be then followed prospectively in the longitudinal cohort study to evaluate end points predictive of cognitive decline and dementia.

The primary objective is: to assess whether retinal sensitivity measured by microperimetry is able to predict cognitive decline and progression to dementia in MCI T2D patients.

The secondary objectives are:

1. To assess whether retinal sensitivity, measured by microperimetry, can identify individuals with MCI among people with T2D.
2. To assess whether eye fixation, measured by microperimetry, can identify individuals with MCI among people with T2D.
3. To assess whether eye fixation measured by microperimetry is able to predict rapid cognitive decline in T2D patients with MCI.
4. To define a T2D phenotype at high risk of developing dementia based on retinal imaging and functional retinal assessments.
5. To determine whether retinal imaging and functional retinal assessments may identify individuals with MCI among people with T2D.
6. To define a T2D phenotype at high risk to develop cognitive decline and dementia based on retinal imaging plus brain imaging.
7. To define a T2D phenotype at high risk to develop dementia based on retinal imaging plus brain imaging plus circulating biomarkers.
8. To establish a score to predict cognitive decline or progression from MCI to dementia based on the variables included in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes
2. 65 years and older
3. Diabetes duration of at least 5 years
4. No overt retinopathy on fundus examination or fundus images, as determined by the evaluating ophthalmologist, in one or both eyes, and people with mild to moderate non-proliferative diabetic retinopathy (NPDR) as determined by the evaluating phthalmologists using fundus examination by slit-lamp biomicroscopy.
5. Able to provide informed consent

Prospective study:

In addition to the above, participants enrolled in the prospective longitudinal cohort study should fulfilled the following criteria:

1. Diagnosis of MCI confirmed by a neuropsychological test battery (NTB) and a specialized physician. For the control group the absence of MCI will also be confirmed by a neuropsychological test battery (NTB) and a specialized physician.
2. Diagnosis of no overt or mild to moderate NPDR (ETDRS DR level 20 to 47) confirmed by the reading centre.

Exclusion Criteria:

1. Previous history of stroke or neurodegenerative diseases.
2. Severe NPDR, Proliferative DR (PDR), Diabetic Macular Edema (DME) or other eye disorders affecting vision besides these complications of diabetic retinopathy (DR).
3. Previous laser photocoagulation.
4. Other diseases which may induce retinal neurodegeneration (e.g. glaucoma).
5. Subjects with a refractive error ≥ ± 6 D.
6. Media opacities that preclude retinal imaging.
7. HbA1C > 10% (86 mmol/mol).
8. Severe systemic illness or personal circumstances that would not make it possible for patients to fulfil study protocols.

Prospective study:

In addition to the above, participants enrolled in the prospective longitudinal cohort study should fulfilled the following criteria:

1. Established dementia.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Subjects with type 2 diabetes, older than 65 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 510 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Retinal sensitivity | 48 month
  Assessed by microperimetry

SECONDARY OUTCOMES:
Retinal neurodysfunction/ neurodegeneration-1 | 48 month
  Assessed by gaze fixation: areas BCEA63, BCEA95 and P1, P2 fixation points will be evaluated
Retinal neurodysfunction/ neurodegeneration-2 | 48 month
  Full-field photopic electroretinogram (ERG)
Retinal neurodysfunction/ neurodegeneration-3 | 48 month
  Spectral Domain Optical Coherence Tomography (SD-OCT): measurement of the retinal layers .
Retinal vascular abnormalities-1 | 48 month
  Assessed by Optical Coherence Tomography Angiography (OCT-A)
Retinal vascular abnormalities-2 | 48 month
  Ultra-wide field Fundus Fluorescein Angiography (FFA).
Brain imaging-1 | 48 month
  Assessed by Magnetic Resonance Imaging (MRI).
Brain imaging-2 | 48 month
  18 Fluoro-2-deoxyglucose-Positron Emission Tomography (18FDG-PET).
Circulating biomarkers: Hypothesis free analysis | 48 month
  Blood samples: proteomics, complement system, inflammatory mediators, glial acidic fibrillary protein, HOMA-IR
Geriatric Depression Scale | 48 month
  Geriatric Depression Scale (GDS-15): scores 0-4 normal, 5-8 mild depression, 9-11 moderate depression, 12-15 severe depression
Quality of life: EQ-5D-3L | 48 month
  EQ-5D-3L questionnaire . The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Visual Functioning Questionnaire | 48 month
  25-item National Eye Institute Visual Functioning Questionnaire (NEI-VFQ-25) . The NEI VFQ-25 contains a reduced number of items within each subscale of the original 51-item NEI VFQ. 13,29 The 12 subscales in the NEI VFQ-25 are general vision, near vision, distance vision, driving, peripheral vision, color vision, ocular pain, general health, and vision-specific role difficulties, dependency, social function, and mental health. The subscale scores are calculated by summing the relevant items and transforming the raw scores into a 0 to 100 scale where higher scores indicate better functioning or well-being. The total score of the NEI VFQ-25 is an average of 11 subscale scores, excluding the single-item general health subscale.
Diabetes Specific Dementia Risk Score. | 48 month
  Diabetes Specific Dementia Risk Score (DSDRS). Briefly,the score is based on the age of the patients, history of any acute metabolic decompensation, the presence micro and/or macrovascular complications of the diabetes, depression and education level, obtaining a score ranged between -1 and 19. The higher the score, more risk of developing dementia at 10 years follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Noemi Lois, Prof., Study Director — Queen´s University Belfast; Rafael Simó, Prof, Study Director — Vall Hebron Research Institute-VHIR
Locations (1):
- Rafael Simó, Barcelona, Spain